CLINICAL TRIAL: NCT03234244
Title: A Randomized, Open-label, Single-dose Study to Evaluate the Safety and the Pharmacokinetics After Oral Concurrent Administration of HDDO-16141 and HDDO-16142 in Healthy Adult Subjects
Brief Title: HDDO-1614 Intervention Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hyundai Pharmaceutical Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: HT-008-01
Record Dates: First submitted 2017-07-26; First posted 2017-07-31 (Actual); Last update posted 2017-12-11 (Actual); Status verified 2017-04

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — bazedoxifene; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bazedoxifene 20mg (Active Comparator): Subjects will take bazedoxifene 1 Tablet.
  Interventions: Drug: Bazedoxifene 20 mg
- Cholecalciferol (Active Comparator): Subjects will take Cholecalciferol 2 Tablets.
  Interventions: Drug: Cholecalciferol
- Bazedoxifene 20mg and Cholecalciferol (Experimental): Subjects will take bazedoxifene 1 tablet and Cholecalciferol 2 tablets at once.
  Interventions: Drug: Bazedoxifene 20mg and Cholecalciferol

INTERVENTIONS:
Drug: Bazedoxifene 20 mg — To estimate the drug-drug interaction between Bazedoxifene and combination of Bazedoxifene and Cholecalciferol, Subject will take Bazedoxifene 20mg 1 tablet one time.
  Arms: Bazedoxifene 20mg
Drug: Cholecalciferol — To estimate the drug-drug interaction between Cholecalciferol and combination of Bazedoxifene and Cholecalciferol, Subject will take Cholecalciferol 2 tablets one time.
  Arms: Cholecalciferol
Drug: Bazedoxifene 20mg and Cholecalciferol — For estimate the Drug-Drug Interaction, Subject will take Bazedoxifene 1 tablet and Cholecalciferol 2 tablets at once.
  Arms: Bazedoxifene 20mg and Cholecalciferol

SUMMARY:
Randomized, Open-label, Single-dose, 3-period, 6-sequence, 3-way crossover Study

ELIGIBILITY:
Inclusion Criteria:

* Body weight 50kg ≤ / BMI=18~29kg/㎡
* A person who is determined to be eligible for the test through a physical examination or an interview
* Those who have been judged to be eligible for the clinical laboratory tests such as hematology test, blood chemistry test, urine test, urine test, serology test

Exclusion Criteria:

* Patients with clinically significant liver, pancreas, kidney, nervous system, respiratory, endocrine, hematologic, mental, cardiovascular
* Patients with a history of gastrointestinal disorders or history of gastrointestinal surgery that may affect the absorption of pharmaceuticals for clinical trials
* Any person who shows any of the following results in the screening test

  1. AST or ALT > 2 times upper limit of normal range
  2. Total Bilirubin > 2.0mg/dL
  3. Glomerular filtration rate (eGFR) < 60mL / min/ 1.7㎡
* Those who show signs of hypotension (systolic blood pressure ≤ 100mmHg or diastolic blood pressure ≤ 55mmHg) or Hypertension (systolic blood pressure ≥ 150mmHg or diastolic blood pressure ≥ 95mmHg)
* Those who have a history of drug abuse or who have a positive urine drug test

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2017-08-14 (Actual); Study Completion 2017-08-14 (Actual)

PRIMARY OUTCOMES:
Drug-Drug Interaction | Day 1~Day 56
  To compare the pharmacokinetic assessment between each comparative drug and combination of bazedoxifene and cholecalciferol.

SECONDARY OUTCOMES:
Pharmacokinetic Assessment | 0, 0.333, 0.667, 1, 1.5, 2, 3, 4, 6, 12, 24, 48, 72, 96 and 120 hours
  Bazedoxifene Maximum Plasma Concentration
Pharmacokinetic Assessment | 0, 0.333, 0.667, 1, 1.5, 2, 3, 4, 6, 12, 24, 48, 72, 96 and 120 hours
  Bazedoxifene Area Under Curve
Pharmacokinetic Assessment | Pre-dose: -24, -18, -12, 0 hour, Post-dose: 2, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48, 72, 96 hour
  Maximun Plasma Concentration after correction of basal concentration of Cholecalciferol
Pharmacokinetic Assessment | Pre-dose: -24, -18, -12, 0 hour, Post-dose: 2, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48, 72, 96 hour
  Area Under Curve after correction of basal concentration of Cholecalciferol

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Heon Cho, Principal Investigator — Inha University Hospital
Locations (1):
- Inha University Hospital, Junggu, Incheon, South Korea